CLINICAL TRIAL: NCT05851430
Title: Galvanize Prospective/Retrospective Pulsed Electric Field Device Registry
Acronym: PROPEL
Status: Recruiting | Type: Observational
Sponsor: Galvanize Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP-00017
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Soft Tissue Lesion
Keywords: Pulsed Electric Fields

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Aliya PEF ablation: Patients will undergo PEF ablation per institutional standard of care
  Interventions: Device: PEF ablation

INTERVENTIONS:
Device: PEF ablation — Pulsed Electric Field (PEF) Ablation per institutional standard of care

SUMMARY:
The goal of this observational registry is to assess the use and performance of Galvanize PEF technology in a real-world setting. The main questions it aims to answer are:

* PEF utilization and performance
* Monitor safety outcomes and inform future generation devices.

Participants will undergo the PEF procedure and be followed per institutional standard of care.

DETAILED DESCRIPTION:
This is a multi-center, observational registry that follows patients for a total of 2 years from the date of the Pulsed Electric Field (PEF) procedure with the FDA cleared Galvanize Technology.

Patients will be enrolled and followed prospectively or enrolled retrospectively with prospective, longitudinal follow up.

Enrollment for this study will include up to 200 patients throughout the US who underwent or are scheduled to undergo PEF energy delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject will undergo or has undergone PEF energy delivery utilizing Galvanize technology
2. Subject is expected to be available for follow-up per the enrolling physician's standard care practices
3. For prospective cohort, subject has a life expectancy of at least 3 months; for retrospective cohort, subject has completed at least three months of imaging following the PEF procedure
4. Signed informed consent is obtained, if required by IRB

Exclusion Criteria:

None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had or who are scheduled to have soft tissue ablated by the Galvanize PEF technology
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Anesthesia Type Usage for PEF Procedure | PEF procedure
  Anesthesia type usage
PEF Target Location | PEF procedure
  PEF procedural target location
PEF Target Size | PEF procedure
  PEF target size (cm)

SECONDARY OUTCOMES:
Incidence of SAEs | within 30 days of PEF energy delivery
  Incidence of SAEs (Registry device and/or procedure related)
Unanticipated [not listed in the Instructions for Use (IFU)] adverse events | within 30 days of PEF energy delivery
  Unanticipated [not listed in the Instructions for Use (IFU)] adverse events (device-related)

CONTACTS AND LOCATIONS:
Overall Officials: William Krimsky, MD, Study Chair — Chief Medical Officer
Locations (4):
- United States (4):
  - Eisenhower Medical Center, Rancho Mirage, California
  - New York Presbyterian Langone Health, New York, New York
  - Duke University Hospital, Durham, North Carolina
  - Lankenau Institute for Medical Research (LIMR), Wynnewood, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
No plan of data sharing